CLINICAL TRIAL: NCT00888784
Title: Endoscopic Cyanoacrylate Injection Versus Beta-Blockers for Secondary Prophylaxis of Gastric Variceal Bleed
Brief Title: Secondary Prophylaxis Gastric Variceal Bleed
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Govind Ballabh Pant Hospital (Other Government)
Responsible Party: Shiv K Sarin, G B Pant Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SRM03
Record Dates: First submitted 2009-04-27; First posted 2009-04-28 (Estimated); Last update posted 2009-04-28 (Estimated); Status verified 2009-04

CONDITIONS: Cirrhosis
MeSH Terms: conditions — Fibrosis | interventions — Adhesives; Adrenergic beta-Antagonists; Propranolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1. Endoscopic Cyanoacrylate injection (Active Comparator): Endoscopic Cyanoacrylate injection in the gastric varix
  Interventions: Procedure: Endoscopic Cyanoacrylate injection
- 2. Beta-blocker (Placebo Comparator): Propranolol was started at a dose of 20 mg twice daily. The principle of incremental dosing was used to achieve the target heart rate for propranolol. The dose was increased every alternate day to achieve a target heart rate of 55/min or to the maximal dose to 360 mg/day if the medication was well tolerated and the systolic blood pressure was >90 mm Hg. On the occurrence of intolerable adverse effects, systolic blood pressure <90 mm Hg or pulse rate <55/min, the dose of the medication was decreased step-wise, and eventually stopped if these adverse events persisted. Reintroduction of the medication was attempted if cessation of the medication did not result in improvement of the reported side-effect.
  Interventions: Drug: beta-blocker (propranolol)

INTERVENTIONS:
Procedure: Endoscopic Cyanoacrylate injection — Endoscopic Cyanoacrylate injection in gastric varix
  Other Names: Glue injection
  Arms: 1. Endoscopic Cyanoacrylate injection
Drug: beta-blocker (propranolol) — Propranolol was started at a dose of 20 mg twice daily. The principle of incremental dosing was used to achieve the target heart rate for propranolol. The dose was increased every alternate day to achieve a target heart rate of 55/min or to the maximal dose to 360 mg/day if the medication was well tolerated and the systolic blood pressure was >90 mm Hg. On the occurrence of intolerable adverse effects, systolic blood pressure <90 mm Hg or pulse rate <55/min, the dose of the medication was decreased step-wise, and eventually stopped if these adverse events persisted. Reintroduction of the medication was attempted if cessation of the medication did not result in improvement of the reported side-effect.
  Arms: 2. Beta-blocker

SUMMARY:
The investigators conducted a randomized, controlled trial (RCT) to study the efficacy of beta blockers versus endoscopic cyanoacrylate injection in the prevention of gastric variceal (GOV2 or IGV1) rebleeding and improvement in survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients with GOV2 without esophageal varix or IGV1, who had bled from GV were included

Exclusion Criteria:

* Presence of esophageal varix
* GOV2 with GOV1; contraindications to beta-blocker therapy and cyanoacrylate injection
* Prior injection of cyanoacrylate or sclerotherapy for GV or GV ligation, transjugular intrahepatic portosystemic shunt, balloon-occluded retrograde transvenous obliteration, balloon-occluded endoscopic injection sclerotherapy of GV, shunt operation for prevention of rebleeding from GV
* Patients already on beta-blocker or nitrates
* Undetermined origin of bleeding from esophageal varix or gastric varix
* Hepatic encephalopathy grade III/IV
* Hepatorenal syndrome
* Hepatocellular carcinoma
* Presence of deep jaundice (serum bilirubin > 10 mg/dl)
* Uremia
* Cerebrovascular accident
* Cardiorespiratory failure
* Pregnancy or patients not giving informed consent for endoscopic procedures

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2006-08; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Rebleeding from GV or death | Overall Study

SECONDARY OUTCOMES:
Increase or decrease in the size of GV, appearance of new esophageal varices and appearance or worsening of portal hypertensive gastropathy and complications. | Overall Study

CONTACTS AND LOCATIONS:
Overall Officials: Shiv K Sarin, MD, DM, Principal Investigator — Director, G B Pant Hospital
Locations (1):
- G B Pant Hospital, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Derived] Mishra SR, Chander Sharma B, Kumar A, Sarin SK. Endoscopic cyanoacrylate injection versus beta-blocker for secondary prophylaxis of gastric variceal bleed: a randomised controlled trial. Gut. 2010 Jun;59(6):729-35. doi: 10.1136/gut.2009.192039. PMID 20551457